CLINICAL TRIAL: NCT01208701
Title: The Effect of Atorvastatin on the NO-system in Patients With Type 2 Diabetes and Nephropathy
Brief Title: The Effects of Atorvastatin on the Nitrogen Oxide-system in Patients With Type 2 Diabetes and Nephropathy
Acronym: STAD
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Erling Bjerregaard Pedersen (Other)
Responsible Party: Sponsor-Investigator, Erling Bjerregaard Pedersen, professor chief physician, Regional Hospital Holstebro
Organization: Regional Hospital Holstebro (Other)
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: EBP-FHC-2010-3
Record Dates: First submitted 2010-09-19; First posted 2010-09-24 (Estimated); Last update posted 2015-08-21 (Estimated); Status verified 2015-08

CONDITIONS: Nephropathy; Cardiovascular Diseases; Diabetes Mellitus
Keywords: Atorvastatin; L-NMMA; NO; Nephrology; Diabetes Mellitus
MeSH Terms: conditions — Kidney Diseases; Cardiovascular Diseases; Diabetes Mellitus | interventions — Atorvastatin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Atorvastatin (Active Comparator)
  Interventions: Drug: Atorvastatin
- Placebo (Placebo Comparator)
  Interventions: Drug: Unikalk

INTERVENTIONS:
Drug: Atorvastatin — Zarator, 80 mg pr day for 5 days
  Other Names: Zarator
  Arms: Atorvastatin
Drug: Unikalk — 1 tablet Unikalk pr day for 5 days
  Arms: Placebo

SUMMARY:
It has been documented that statin reduce mortality and morbidity in patients with cardiovascular disease. This effect can partly be related to a reduction in cholesterol levels in blood. Nitric oxide (NO) production is reduced in several chronic diseases such as nephropathy, diabetes and hypertension. The purpose of this study is to investigate the effect of Atorvastatin treatment on the NO-system measuring renal and cardiovascular variables in patients with type 2 diabetes with nephropathy.

DETAILED DESCRIPTION:
Subjects will be examined on two examination days. 4 days prior to each examination day subjects are treated with either atorvastatin or placebo. During treatment periods subject are given a standardized diet.

On the examination days subject are given L-NMMA(L-NG-monomethyl Arginine citrate), a NO inhibitor, 6 mg bolus infusion followed by continuous 4 mg/kg/hr infusion for 1 hour. Renal function, central hemodynamic and vasoactive hormones are evaluated prior, during and after L-NMMA infusion.

Renal function is measured by renal clearance of 51Cr-EDTA and urinary sodium, potassium and albumin concentration. Urinary excretion of protein from sodium channels such as the NaCl cotransporter (NCC), the Na-K-Cl cotransporter (NKCC) and the epithelial sodium channel (ENaC) will be measured to evaluate channel activity in the nephron.

Central blood pressure, pulse wave analysis, and augmentation index are measured using SphygmoCor® from Atcor.

ELIGIBILITY:
Inclusion Criteria:

* Men and women
* minimum 40 years
* Chronic Kidney disease
* Estimated GFR (eGFR) between 30 and 90 ml/min
* Diabetes Mellitus type II

Exclusion Criteria:

* Nephrotic Syndrome
* Anamnestic or clinical signs of significant heart, lung, lever, kidney and brain disease
* Neoplastic disease
* Alcohol abuse,
* Drug abuse
* Pregnancy or nursing
* Blood donation within a month before examination
* Hgb < 6,0

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2010-05; Primary Completion 2012-01 (Actual); Study Completion 2012-01 (Actual)

PRIMARY OUTCOMES:
Fractional excretion of sodium | 5 days treatment

SECONDARY OUTCOMES:
Systolic blood pressure | 5 days
Plasma renin concentration | 5 days
Arterial stiffness | 5 days
Plasma angiotensin II concentration | 5 days
Urinary excretion of protein from sodium channels such as the NaCl cotransporter (NCC), the Na-K-Cl cotransporter (NKCC) and the epithelial sodium channel (ENaC) | 5 days
Augmentations index | 5 days

CONTACTS AND LOCATIONS:
Overall Officials: Frank H Christensen, MD, Principal Investigator — Department of Medical Research
Locations (1):
- Medicinsk Forskning, Regionshospitalet Holstebro, Holstebro, Denmark

REFERENCES:
- [Derived] Tunnicliffe DJ, Palmer SC, Cashmore BA, Saglimbene VM, Krishnasamy R, Lambert K, Johnson DW, Craig JC, Strippoli GF. HMG CoA reductase inhibitors (statins) for people with chronic kidney disease not requiring dialysis. Cochrane Database Syst Rev. 2023 Nov 29;11(11):CD007784. doi: 10.1002/14651858.CD007784.pub3. PMID 38018702
- [Derived] Mose FH, Larsen T, Jensen JM, Hansen AB, Bech JN, Pedersen EB. Effect of atorvastatin on renal NO availability and tubular function in patients with stage II-III chronic kidney disease and type 2 diabetes. Scand J Clin Lab Invest. 2014 Jan;74(1):8-19. doi: 10.3109/00365513.2013.855942. Epub 2013 Nov 21. PMID 24256611